CLINICAL TRIAL: NCT07313384
Title: Dietary Insights and Nutrition Experiences in Adults on GLP-1 Therapy - A Study on Diet Quality Changes in Adults on GLP-1 Therapy
Acronym: DINE-GLP1
Status: Recruiting | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Shiba Simon Bailey, Posdoctoral Fellow, University of South Carolina
Other Study IDs: 2371702-1
Record Dates: First submitted 2025-12-01; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Obesity Type 2 Diabetes Mellitus; Obesity (Disorder)
Keywords: GLP-1 Therapy; Nutrition Support; Obesity; Weight loss therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLP-1 Therapy: Individuals prescribed with GLP-1 Therapy for obesity or T2DM management.
  Interventions: Drug: GLP-1 Therapy

INTERVENTIONS:
Drug: GLP-1 Therapy — Exposure to GLP-1 Therapy for obesity or T2DM management.

SUMMARY:
The DINE-GLP1 study aims to understand how people on GLP-1 therapy change their eating habits and what kind of dietary support they need. As more people use GLP-1 medications, there's not much guidance on what they should eat, mostly just focusing on managing symptoms and cutting calories. Since these medications reduce food intake, it's important to ensure the diet is nutritious even with fewer calories to help with long-term weight control and health. Most research has looked at how the body responds to the medication and whether patients take it as prescribed, but not much is known about what patients actually experience, what they think they need, or how they could use additional support. Understanding patients' views can help create better lasting solutions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Recently has been prescribed GLP-1 therapy for the treatment of obesity or T2DM but have not yet initiated the medication
* Has regular access to a smartphone and internet to complete short surveys and food recalls online
* Willing to sign informed consent.

Exclusion Criteria:

* Already began the GLP-1 medication
* Have medical concerns making participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will be conducted at the Prisma Health Weight Management Institute in Greenville, South Carolina, with support from the on-site research team. A total of 50 patients will be enrolled. Eligible individuals will be adults aged 18 years or older who have recently been prescribed GLP-1 therapy for the treatment of obesity or T2DM but have not yet initiated the medication.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Eating Index | Baseline and 12-weeks
  The Healthy Eating Index (HEI) is a scoring metric developed by the U.S. Department of Agriculture (USDA) and the NCI to assess how well a person's diet conforms to the Dietary Guidelines for Americans. It evaluates the consumption of 13 dietary components, including both adequacy (foods to increase) and moderation (foods to decrease). The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations and dietary patterns published in the Dietary Guidelines.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline and 12 weeks
  Change from Baseline in Body Weight at 12-weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University South Carolina, Columbia, South Carolina
  - Prisma Health Weight Management Institute, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided